CLINICAL TRIAL: NCT04976543
Title: Initiation of NWS Anticoagulation Therapy After Oesophageal Variceal Band Ligation Was Safe in Portal Vein Thrombosis Patients With Cirrhosis and Acute Variceal Bleeding: A Multi-central Randomized Controlled Trial
Brief Title: Safety of Anticoagulant Therapy After Endoscopic Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Qilu Hospital of Shandong University (Other)
Collaborators: Liaocheng People's Hospital (Other); Taian City Central Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20200202-Qilu
Record Dates: First submitted 2021-07-15; First posted 2021-07-26 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2020-02

CONDITIONS: Cirrhosis; Portal Vein Thrombosis; Esophageal and Gastric Varices; Anticoagulant-induced Bleeding
Keywords: endoscopic therapy; endoscopic variceal band ligation; warfarin; nadroparin calcium
MeSH Terms: conditions — Fibrosis; Esophageal and Gastric Varices

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NWS group (Experimental): nadroparin calcium injection subcutaneously every 12 hours for 1 month and switched to warfarin orally for 5 months
  Interventions: Drug: nadroparin calcium-warfarin sequential anticoagulation
- control group (No Intervention): no anticoagulation therapy

INTERVENTIONS:
Drug: nadroparin calcium-warfarin sequential anticoagulation — The NWS therapy group were given a subcutaneous injection of nadroparin calcium every 12 hours for 1 month and switched to warfarin for 5 months. Warfarin was initiated at least 5 days before nadroparin calcium was stopped. International normalized ratio (INR) was detected every 3-4 days and adjusted carefully by 0.75mg dosage until achieve the target level of 2-3.
  Other Names: anticoagulation
  Arms: NWS group

SUMMARY:
The investigators aimed to verify the efficacy and safety of nadroparin calcium warfarin sequential (NWS) anticoagulation therapy after endoscopic therapy in PVT patients with cirrhosis and AVB.

DETAILED DESCRIPTION:
Acute variceal bleeding is one of the most serious complications of liver cirrhosis and is associated with significant morbidity and mortality. Portal vein thrombosis (PVT) aggravates portal hypertension and worsens hemorrhage, which Increases the risk of endoscopic therapy, and PVT has been shown to be associated with a longer time to variceal eradication, a higher risk of variceal relapse and rebleeding. So, PVT should be treated earlier. Data regarding the safety and initiation time of anticoagulant therapy in PVT patients with variceal bleeding after endoscopic therapy is lacking. Aim of this study is to verify the efficacy and safety of NWS anticoagulation therapy in PVT patients with cirrhosis and AVB after endoscopic therapy and further to explored the appropriate initiation time of NWS anticoagulation therapy after EVL in these patients.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of cirrhosis
* Portal hypertension with esophageal and gastric varices
* diagnosis of PVT by imaging examination
* undergo endoscopic therapy

Exclusion Criteria:

* older than 75 years
* uncontrolled active bleeding
* hepatocellular carcinoma or other extrahepatic malignancy
* on-going or received antithrombotic/thrombolytic treatment
* previous treatment with TIPSS
* cavernous transformation of the portal vein
* platelet count lower than 10*10 ^ 9/L, creatinine more than 170 μmol/L
* Budd-Chiari syndrome
* pregnancy or breast-feeding period
* severe cardiopulmonary diseases, severe systemic infection or sepsis
* inability to sign informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-06-28 (Actual)

PRIMARY OUTCOMES:
rate of overall recanalization | 6-month
  the sum of the fraction of patients who had complete or partial recanalization
rate of bleeding | 6-month
  rates of upper gastrointestinal (GI) rebleeding, epistaxis, injection-site hemorrhage, and other bleeding events

CONTACTS AND LOCATIONS:
Overall Officials: Yanjing Gao, PhD.MD, Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Department of Gastroenterology,Qilu Hospital,Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No